CLINICAL TRIAL: NCT00628394
Title: Cognitive Treatments in Schizophrenia
Brief Title: Treating Cognition in Schizophrenia With Atomoxetine and Cognitive Remediation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Carol A. Tamminga, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0803-476; 1R34MH075863-01A2 (NIH)
Record Dates: First submitted 2008-02-24; First posted 2008-03-05 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Cognition in Schizophrenia
Keywords: Cognition; schizophrenia; Atomoxetine; Strattera; cognitive remediation
MeSH Terms: conditions — Schizophrenia | interventions — Atomoxetine Hydrochloride; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Atomox/CR (Other): Patients are given the drug Atomoxetine and Cognitive Remediation training.
  Interventions: Drug: Atomoxetine
- Atomox/Control (Other): Patients are given the drug Atomoxetine and Remediation Control training.
  Interventions: Drug: Atomoxetine
- Placebo/CR (Other): Patients are given a Placebo and Cognitive Remediation training.
  Interventions: Drug: Placebo
- Placebo/Control (Other): Patients are given Placebo and Remediation Control training.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — 40mg 2po qam
  Other Names: Strattera
  Arms: Atomox/CR; Atomox/Control
Drug: Placebo — 40mg 2po qam
  Other Names: Cornstarch capsule
  Arms: Placebo/CR; Placebo/Control

SUMMARY:
This research is being done because people with schizophrenia often have problems with thinking including learning, remembering, paying attention, and problem solving. During this study, we will test if cognitive remediation (computer games made to improve thinking), used along with a drug called atomoxetine, may help the problems in thinking as well as some of the symptoms of schizophrenia.

DETAILED DESCRIPTION:
Persons with schizophrenia in a stable and residual antipsychotic- treated clinical condition for at least 8 weeks will be recruited from several public mental health treatment settings into the UTSW Schizophrenia Research Clinic. Each volunteer will receive information about the protocol and its risks and benefits. If they give their informed consent after a full opportunity to learn about the details of the study, they will be allowed to proceed. All recruits will have been treated with optimal dosing of any 2nd generation antipsychotic drug (APD-2) and will have been clinically stable with respect to psychotic symptoms for at least 6 weeks prior to randomization, and on a stable dose of the medication for at least 2 weeks. All eligible volunteers will receive a routine medical assessment and psychiatric diagnostic work-up including the SCID and a consensus diagnosis by two experienced clinicians based on all available data, prior to the randomization. Just prior to randomization, the following sets of assessments will be performed: (1) Medical: Physical Examination, Clinical Chemistries, EKG, urinalysis, weight, and vital signs; (2) Symptomatic: general psychiatric symptom assessment, including the scores on the PANSS, Psychosis Change Scale, and CGI; (3) Cognitive: standard neuropsychometric test battery and surrogate psychosocial tests; all of the assessment batteries will be repeated at the end of the 12-week treatment period, and repeated again at the end of the three month follow-up period (at 6 months from study start). Clinical symptom scales, weight, and vital signs will be repeated at weeks 4, 8, 12, 16 , and 24 during the study.

The schizophrenia volunteers will be randomized into four treatment groups: (1) atomoxetine plus cognitive remediation; (2) atomoxetine plus remediation control; (3) placebo plus cognitive remediation; and (4) placebo plus remediation control. Atomoxetine or matching placebo will be administered at a dose of 40mg bid (80mg/day) or the placebo equivalent. The remediation sequence will last for 60 minutes and will be administered three times weekly; the remediation control will be administered on the same schedule and for the same duration. Because the volunteers attend the clinic so regularly, we will have an opportunity to track their progress, monitor medication adherence, and optimize study participation.

Then, each volunteer will be followed up while taking their blinded study medications, but without any more remediation/control sessions, for the next 3 months. Psychiatric rating scales will be completed the following times, relative to the blinded randomization: baseline, 1, 2, 3, 4, 5, 6 months, whereas the neuropsychological battery will be completed at baseline and at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder.
* Males and females.
* Ages 18-60 years old.
* All races and ethnicities.

Exclusion Criteria:

* Diagnosis of an organic brain disease.
* Diagnosis of DSM-IV alcohol or substance abuse within the last month or DSM-IV alcohol or substance dependence within the last 3 months.
* Meet criteria for primary negative symptoms, established by clinical judgment.
* Current or past history of clozapine treatment for antipsychotic non-response.
* Patients hospitalized in a psychiatric hospital within the previous 30 days.
* Patients with an unstable medical condition, as determined by the Investigator
* Colorblindness
* Concurrent treatment with electroconvulsive therapy or psychotherapy.
* Pregnant women.
* Must be able to read, speak, and understand English.

  * We do not have the resources necessary to properly study non-English speaking patients in this study. The computer software used for cognitive remediation and some clinical assessments are only available in English. The need to provide such resources in foreign languages would be prohibitive to the successful completion of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2003-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Tamminga, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some participants were never randomized due to Screening labs, illicit substances (repeatedly - exclusion), transportation issues, or simply being lost to follow-up. Lost to f/u were contacted 3 times and sent a letter in order to bring them back into the study.
Period: Overall Study
Arm/Group | Atomox/CR | Atomox/Control | Placebo/CR | Placebo/Control
Started (Participants that made it past Randomization and one session of CR/Control.) | 14 | 13 | 13 | 13
Completed | 10 | 9 | 11 | 10
Not Completed | 4 | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomox/CR | Atomox/Control | Placebo/CR | Placebo/Control | Total
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 11 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 7 | 8 | 29
  Male | 2 | 3 | 4 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 9 | 9 | 11 | 9 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 7 | 5 | 17
  White | 7 | 7 | 4 | 5 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 11 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychological Measures for MATRICS
Description: Gordon Continuous Performance Test - Distractibility Version The test is designed assess a person's executive functioning by testing their ability to maintain their focus over a period of time. They are intended to respond to a series of targets or inhibit their responses to a variety of foils. They are mainly assessed for their omissions and commissions. The omission and commission errors assess the person's ability to screen out extraneous stimuli while responding correctly and inhibiting incorrect responding. This means lower scores are better. The scale is 0-126.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Atomox/CR | Atomox/Control | Placebo/CR | Placebo/Control
Number analyzed (Participants) | 10 | 9 | 11 | 10
score on a scale | 20.82 (1.71) | 18.03 (1.77) | 25.43 (1.64) | 11.64 (1.70)

2. Secondary Outcome: Clinical Outcomes
Description: Birchwood Social Function Scale (SFS) This scale is given to determine a person's ability to function independently and in social settings without difficulty. It assesses a variety of settings with independent subscales (whose scores vary in range) but in which the higher score is always better. These subscales (Withdrawal/Social Engagement; Interpersonal Communication; Independence-Performance; Independence-Competence; Recreation; Prosocial; and, Employment/Occupation) are combined and developed into a mean score. These scores range from 0-32.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomox/CR | Atomox/Control | Placebo/CR | Placebo/Control
Number analyzed (Participants) | 10 | 9 | 11 | 10
units on a scale | 9.75 (.37) | 10.32 (.39) | 10.82 (.36) | 9.02 (.38)

ADVERSE EVENTS:
Arm/Group | Atomox/CR | Atomox/Control | Placebo/CR | Placebo/Control
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 2/9 | 0/11 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomox/CR (N=10) | Atomox/Control (N=9) | Placebo/CR (N=11) | Placebo/Control (N=10)
Decreased appetite (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No